CLINICAL TRIAL: NCT04085822
Title: A Histologic Study of Silk Medical Aesthetics Device in the Abdomen of Patients Undergoing Abdominoplasty
Brief Title: Histology of SMA-001 in the Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silk Medical Aesthetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN-DF-001
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Abdominoplasty; Medical Aesthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Multiple Abdominal Injections (Experimental): Ten injections per patient: 7 of SMA-001 and 3 of control device.
  Interventions: Device: SMA-001

INTERVENTIONS:
Device: SMA-001 — Intra-dermal injection of SMA-001 and control device.

SUMMARY:
Silk Medical Aesthetics' Inc. device, SMA-001, is currently under development as a dermal filler to fill wrinkles and folds. This study is designed to collect short-term visual, photographic, and histological and safety data on small aliquots of the product as part of device development. It is an open label study involving up to three investigational sites and a maximum enrollment of 10 subjects. Juvéderm Ultra Plus XC, an FDA-approved dermal filler will serve as a control device. Briefly, the investigational product and the control device will be injected into the abdomen of patients intending to undergo abdominoplasty at a later date. The patients will be followed for 30 days post injection through visual observation. At 30 days post injection, the injected gel and associated tissue will be removed via biopsy during the abdominoplasty surgery and histology slides created for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 25-65 years of age
2. Abdominoplasty patients with sufficient skin quality (dermal thickness & integrity, limited stretch marks/attenuated skin)
3. Able to follow study instructions and likely to complete all required visits, as assessed by the PI
4. Signed the IRB-approved Informed Consent form and the HIPAA form prior to performance of any study-related procedures

Exclusion Criteria:

1. Subjects with intrinsic skin disease or documented dermatologic conditions
2. Subjects with known bleeding disorders or on medications that may interfere with bleeding
3. Subjects currently taking immunosuppressive drugs, steroids, or anti-inflammatories
4. Subjects receiving injection of lipolytic drugs
5. Subjects with a history of keloid formation or hypertrophic scarring
6. Subjects with documented Type I or II Diabetes Mellitus.
7. Inability or unwillingness of the subject to complete the clinical protocol as described in the protocol and allow access to clinical records.
8. Subjects who are known to be pregnant at the time of enrollment or plan to become pregnant in the coming 30 days.
9. Subjects with documented active drug or alcohol abuse within the last 12 months prior to the study.
10. Subjects with systemic collagen disorders, such as Ehlers Danlos.
11. Subjects with known allergies to hyaluronic acid, silk, lidocaine, and/or Polyethylene Glycol.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Histological performance | 4 weeks
  Four week histology data

SECONDARY OUTCOMES:
Safety | 4 weeks
  Safety of the device through Adverse Event tracking

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Skincare Physicians, Inc, Chestnut Hill, Massachusetts
  - Gryskiewicz Twin Cities Cosmetic Surgery, Burnsville, Minnesota
  - Jewell Plastic Surgery, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No